CLINICAL TRIAL: NCT02354885
Title: Administration of Tranexamic Acid in the Preclinical Setting and Its Effect on Coagulation Parameters and Outcome in Multiple Trauma Patients and Isolated TBI in EMS (Schutz Und Rettung Zürich) and Helicopter Rescue(REGA).
Brief Title: TXA in the EMS on the Helicopter and the Ambulance
Acronym: TXASRZREGA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Oliver Theusinger, PD Dr med, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2014-0069
Record Dates: First submitted 2015-01-16; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tranexamic Acid (No Intervention): TXA administered to multiple trauma patients in the helicopter or ambulance
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Coagulation Management / Efficiency
  Other Names: ROTEM

SUMMARY:
Coagulopathy in trauma increases mortality and morbidity. Early administration of tranexamic acid (TXA) seems to improve survival and outcome. Thus this study evaluates the administration of TXA on scene by the emergency medical services (EMS) or by the crew of a rescue helicopter in multiple trauma patients or isolated traumatic brain injury (TBI). Coagulopathy will be assessed by standard laboratory tests as well as thromboelastometry.

DETAILED DESCRIPTION:
Coagulopathy in trauma increases mortality and morbidity. Early administration of tranexamic acid (TXA) seems to improve survival and outcome; this was shown partially by the CRASH2 study, where patients received TXA in the emergency room. Thus this study evaluates the administration of TXA on scene by the EMS or by the crew of a rescue helicopter in multiple trauma patients or isolated TBI. Coagulopathy will be assessed by standard laboratory tests as well as thromboelastometry in 50 patients. The results will be compared to a study published by Theusinger et al. (Changes in Coagulation in Standard Laboratory Tests and ROTEM in Trauma Patients Between On-Scene and Arrival in the Emergency Department.Theusinger OM et al. Anesth Analg. 2014 Dec 24. [Epub ahead of print] PMID: 25545751) where no TXA was administered on scene and only changes in coagulation between on scene and in the emergency department were assessed.

ELIGIBILITY:
Inclusion Criteria:

* multiple trauma
* traumatic brain injury

Exclusion Criteria:

* pregnant
* < 18 years
* no TXA
* not speaking the german language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Tranexamic acid administered in the preclinical setting and its influence on coagulation parameters (laboratory and thromboelastometry) | 12 Months
  TXA will be given to multiple trauma patients or patients with isolated TBI in the preclinical setting (n=50). Before tranexamic acid is given, one tube of citrated blood is drawn. Once patients arrive in the emergency room as second tube of citrated blood is drawn. The two tubes will be used to perform rotational thromboelastometry (ROTEM) measurements and standard coagulation measurements (aPTT, PT, INR, Ouick's value, fibrinogen). The coagulation parameters on scene will be compared to those in the emergency department to find out if coagulation is improved by this. In a previously performed study, 50 patients got blood taken on scene and in the emergency room without receiving TXA. In this study by Theusinger et al. it was shown that coagulation is impaired during this time period.(Theusinger OM et al. Anesth Analg. 2014 Dec 24.PMID: 25545751). The population of this study will serve as control group for the actually performed study.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver M. Theusinger, PD Dr med, Principal Investigator — USZ
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Division of Anaesthesiology, Zurich, Canton of Zurich
  - USZ, Zurich

REFERENCES:
- [Derived] Stein P, Studt JD, Albrecht R, Muller S, von Ow D, Fischer S, Seifert B, Mariotti S, Spahn DR, Theusinger OM. The Impact of Prehospital Tranexamic Acid on Blood Coagulation in Trauma Patients. Anesth Analg. 2018 Feb;126(2):522-529. doi: 10.1213/ANE.0000000000002708. PMID 29239953